CLINICAL TRIAL: NCT03191110
Title: The COLON Study: Colorectal Cancer: Longitudinal, Observational Study on Nutritional and Lifestyle Factors That May Influence Colorectal Tumour Recurrence, Survival and Quality of Life
Brief Title: The COLON Study: Colorectal Cancer Cohort
Acronym: COLON
Status: Active, not recruiting | Type: Observational
Sponsor: Wageningen University (Other)
Collaborators: Dutch Cancer Society (Other); Wereld Kanker Onderzoek Fonds (Other); Funding: World Cancer Research Fund International (Unknown); Funding: ERA-NET on Translational Cancer Research (TRANSCAN) (Unknown)
Responsible Party: Principal Investigator, Ellen Kampman, prof. dr. ir. Ellen Kampman, Wageningen University
Other Study IDs: NL30446.091.09; CMO number 2009/349 (Other: Medical Ethical Committee)
Record Dates: First submitted 2017-06-09; First posted 2017-06-19 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Neoplasms Malignant
Keywords: COLON; colorectal cancer; nutrition; lifestyle; survival; recurrence; quality of life
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for all participants. Stool samples will be collected in a subgroup of colon cancer patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Colorectal cancer patients
  Interventions: Other: No intervention: observational study

INTERVENTIONS:
Other: No intervention: observational study

SUMMARY:
The main aim of this observational, prospective cohort study is to assess associations of diet and other lifestyle factors with colorectal cancer recurrence, survival and quality of life.

DETAILED DESCRIPTION:
The COLON study is a multi-centre prospective cohort study among incident colorectal cancer patients recruited from 12 hospitals in the Netherlands. Patients with colorectal cancer are invited upon diagnosis. Upon recruitment, after 6 months, 2 years and 5 years, patients fill out food-frequency questionnaires; questionnaires about dietary supplement use, physical activity, weight, height, and quality of life; and donate blood samples. Diagnostic CT-scans are collected to assess cross-sectional areas of skeletal muscle, subcutaneous fat, visceral fat and intermuscular fat, and to assess muscle attenuation. Blood samples are biobanked to facilitate future analyse of biomarkers, nutrients, DNA etc. Analysis of serum 25-hydroxy vitamin D levels, B-vitamins and metabolomic profiles are scheduled. A subgroup of patients with colon cancer is asked to provide faecal samples before and at several time points after colon resection to study changes in gut microbiota during treatment. For all patients, information on vital status is retrieved by linkage with national registries. Information on clinical characteristics, including treatment-related toxicity and co-morbidity data, is gathered from linkage with the Netherlands Cancer Registry and with hospital databases or medical records. Hazard ratios will be calculated for dietary and lifestyle factors at diagnosis in relation to recurrence and survival. Repeated measures analyses will be performed to assess changes over time in dietary and other factors in relation to recurrence and survival.

The aim is to recruit at least 2000 patients with available data and blood samples.

ELIGIBILITY:
Inclusion Criteria:

- Patients newly diagnosed with colorectal cancer in one of the participating hospitals

Exclusion Criteria:

* Non-Dutch speaking
* A history of colorectal cancer or (partial) bowel resection
* Chronic inflammatory bowel disease
* Hereditary colorectal cancer syndromes (Lynch syndrome, FAP, Peutz-Jegher)
* Dementia or another mental condition that makes it impossible to fill out questionnaires

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men and women of all ages, who were newly diagnosed with colorectal cancer (ICD codes C18-20) in any stage of the disease in one of the participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-08-03 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Survival | An average follow-up of at least 5 years
  Overall survival
Cancer recurrence | An average follow-up of at least 5 years
  Cancer recurrence
Quality of life (EORTC QLQ-C30) | An average follow-up of at least 5 years
  Quality of life

SECONDARY OUTCOMES:
Chemotherapy-induced toxicity (QLQ-CIPN20) | 12 months after diagnosis
  Chemotherapy-induced peripheral neuropathy
Microbiota composition based on 16S rRNA profiling | At diagnosis and 6, 12 and 35 weeks after resection
  Stool samples
Co-morbidities | An average follow-up of at least 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Kampman, PhD, Principal Investigator — Wageningen University
Locations (11):
- Netherlands (11):
  - Ziekenhuisgroep Twente, Almelo
  - Gelre Hospital, Apeldoorn
  - Rijnstate Hospital, Arnhem
  - Slingeland Hospital, Doetinchem
  - Hospital Gelderse Vallei, Ede
  - Admiraal De Ruyter Hospital, Goes/Vlissingen
  - Martini Hospital, Groningen
  - Canisius Wilhelmina Hospital, Nijmegen
  - Radboudumc, Nijmegen
  - Bernhoven Hospital, Oss
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Winkels RM, Heine-Broring RC, van Zutphen M, van Harten-Gerritsen S, Kok DE, van Duijnhoven FJ, Kampman E. The COLON study: Colorectal cancer: Longitudinal, Observational study on Nutritional and lifestyle factors that may influence colorectal tumour recurrence, survival and quality of life. BMC Cancer. 2014 May 27;14:374. doi: 10.1186/1471-2407-14-374. PMID 24886284
- [Derived] Klaassen-Dekker N, Zoetendal EG, Capuano E, Winkels RM, van Duijnhoven FJ, van Heek NT, Kruyt FM, Ulvik A, McCann A, Ueland PM, de Wilt JH, Kampman E, Kok DE. Preoperative plasma short- and branched-chain fatty acids in relation to risk of complications after colorectal cancer surgery: a prospective cohort study. Am J Clin Nutr. 2025 Dec;122(6):1579-1590. doi: 10.1016/j.ajcnut.2025.10.001. Epub 2025 Oct 10. PMID 41076267
- [Derived] Smit KC, Derksen JWG, Stellato RK, VAN Lanen AS, Wesselink E, Belt EJT, Balen MC, Coene PPLO, Dekker JWT, DE Groot JW, Haringhuizen AW, VAN Halteren HK, VAN Heek TT, Helgason HH, Hendriks MP, DE Hingh IHJT, Hoekstra R, Houtsma D, Janssen JJB, Kok N, Konsten JLM, Los M, Meijerink MR, Mekenkamp LJM, Peeters KCMJ, Polee MB, Rietbroek RC, Schiphorst AHW, Schrauwen RWM, Schreinemakers J, Sie MPS, Simkens L, Sonneveld EJA, Terheggen F, Iersel LV, Vles WJ, Wasowicz-Kemps DK, DE Wilt JHW, Kok DE, Winkels RM, Kampman E, VAN Duijnhoven FJB, Koopman M, May AM. Determinants of Physical Activity among Patients with Colorectal Cancer: From Diagnosis to 5 Years after Diagnosis. Med Sci Sports Exerc. 2024 Apr 1;56(4):623-634. doi: 10.1249/MSS.0000000000003351. Epub 2023 Nov 27. PMID 38079324
- [Derived] Kok DE, van Duijnhoven FJ, Lubberman FJ, McKay JA, Lanen AV, Winkels RM, Wesselink E, van Halteren HK, de Wilt JH, Ulrich CM, Ulvik A, Ueland PM, Kampman E. Intake and biomarkers of folate and folic acid as determinants of chemotherapy-induced toxicities in patients with colorectal cancer: a cohort study. Am J Clin Nutr. 2024 Feb;119(2):294-301. doi: 10.1016/j.ajcnut.2023.11.023. Epub 2023 Dec 7. PMID 38070682
- [Derived] van Lanen AS, Kok DE, Wesselink E, Winkels RM, van Halteren HK, de Wilt JHW, Kampman E, van Duijnhoven FJB. Pre- and post-diagnostic dairy intake in relation to recurrence and all-cause mortality in people with stage I-III colorectal cancer. Eur J Nutr. 2023 Oct;62(7):2891-2904. doi: 10.1007/s00394-023-03201-0. Epub 2023 Jul 2. PMID 37393586
- [Derived] Wesselink E, Valk AW, Kok DE, Lanen AV, de Wilt JH, van Kouwenhoven EA, Schrauwen RW, van Halteren HK, Winkels RM, Balvers MG, Kampman E, van Duijnhoven FJ. Postdiagnostic intake of a more proinflammatory diet is associated with a higher risk of recurrence and all-cause mortality in colorectal cancer survivors. Am J Clin Nutr. 2023 Feb;117(2):243-251. doi: 10.1016/j.ajcnut.2022.11.018. Epub 2022 Dec 22. PMID 36811565
- [Derived] Geijsen AJMR, Kok DE, van Zutphen M, Keski-Rahkonen P, Achaintre D, Gicquiau A, Gsur A, Kruyt FM, Ulrich CM, Weijenberg MP, de Wilt JHW, Wesselink E, Scalbert A, Kampman E, van Duijnhoven FJB. Diet quality indices and dietary patterns are associated with plasma metabolites in colorectal cancer patients. Eur J Nutr. 2021 Sep;60(6):3171-3184. doi: 10.1007/s00394-021-02488-1. Epub 2021 Feb 5. PMID 33544207
- [Derived] Wesselink E, Kok DE, de Wilt JHW, Bours MJL, van Zutphen M, Keulen ETP, Kruyt FM, Breukink SO, Kouwenhoven EA, van den Ouweland J, Weijenberg MP, Kampman E, van Duijnhoven FJB. Sufficient 25-Hydroxyvitamin D Levels 2 Years after Colorectal Cancer Diagnosis are Associated with a Lower Risk of All-cause Mortality. Cancer Epidemiol Biomarkers Prev. 2021 Apr;30(4):765-773. doi: 10.1158/1055-9965.EPI-20-1388. Epub 2021 Feb 2. PMID 33531437
- [Derived] Wesselink E, Staritsky LE, van Zutphen M, Geijsen AJMR, Kok DE, Kruyt F, Veenstra RP, Spillenaar Bilgen EJ, Kouwenhoven EA, de Wilt JHW, Kampman E, van Duijnhoven FJB. The association between the adapted dietary inflammatory index and colorectal cancer recurrence and all-cause mortality. Clin Nutr. 2021 Jun;40(6):4436-4443. doi: 10.1016/j.clnu.2021.01.004. Epub 2021 Jan 11. PMID 33478795
- [Derived] van Baar H, Bours MJL, Beijer S, van Zutphen M, van Duijnhoven FJB, Kok DE, Wesselink E, de Wilt JHW, Kampman E, Winkels RM. Body composition and its association with fatigue in the first 2 years after colorectal cancer diagnosis. J Cancer Surviv. 2021 Aug;15(4):597-606. doi: 10.1007/s11764-020-00953-0. Epub 2020 Oct 17. PMID 33067775
- [Derived] Wesselink E, Kok DE, Bours MJL, de Wilt JHW, van Baar H, van Zutphen M, Geijsen AMJR, Keulen ETP, Hansson BME, van den Ouweland J, Witkamp RF, Weijenberg MP, Kampman E, van Duijnhoven FJB. Vitamin D, magnesium, calcium, and their interaction in relation to colorectal cancer recurrence and all-cause mortality. Am J Clin Nutr. 2020 May 1;111(5):1007-1017. doi: 10.1093/ajcn/nqaa049. PMID 32190892
- [Derived] Wesselink E, Bours MJL, de Wilt JHW, Aquarius M, Breukink SO, Hansson B, Keulen ETP, Kok DE, van den Ouweland J, van Roekel EH, Snellen M, Winkels R, Witkamp RF, van Zutphen M, Weijenberg MP, Kampman E, van Duijnhoven FJB. Chemotherapy and vitamin D supplement use are determinants of serum 25-hydroxyvitamin D levels during the first six months after colorectal cancer diagnosis. J Steroid Biochem Mol Biol. 2020 May;199:105577. doi: 10.1016/j.jsbmb.2020.105577. Epub 2020 Jan 7. PMID 31917319
- See also: Website for studies on Diet and Cancer, Division of Human Nutrition, Wageningen University — http://www.colon-studie.nl/colonstudy_eng